CLINICAL TRIAL: NCT05651113
Title: Exploring Parents' and Health Professionals' Experiences of Screening for Severe Combined Immunodeficiency
Brief Title: The Experience of Screening for SCID
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: University of Manchester (Other); University of Sheffield (Other); Coventry University (Other); National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Jane Chudleigh, Principal Investigator, King's College London
Other Study IDs: SCID Protocol 5Aug2022 V4
Record Dates: First submitted 2022-11-29; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Severe Combined Immunodeficiency
MeSH Terms: conditions — Severe Combined Immunodeficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Positive NBS for SCID: Parents whose baby was referred to an immunologist due their SCID screening result (minimum n= 10-25)
  Interventions: Other: SCID Screening
- Normal NBS result: Parents who received a normal screening result (minimum n=10-25)
  Interventions: Other: SCID Screening
- False positive NBS result: Parents who have received a false positive result elsewhere in screening (minimum n=2-10)
- CFSPID Designation: Parents who received a CFSPID result (minimum n=~10)
- SCID via family history or clinical presentation: Parents whose baby was identified with SCID due to family history or clinical presentation (minimum n=10)
- Parents whose babies have died: Parents who have received an abnormal screening result (T cell receptor excision circles (TRECs) or who were identified with SCID due to family history or clinical presentation and whose baby has subsequently died (n=~10)
  Interventions: Other: SCID Screening

INTERVENTIONS:
Other: SCID Screening — The addition of newborn bloodspot screening for severe combined immunodeficiency
  Groups: Normal NBS result; Parents whose babies have died; Positive NBS for SCID

SUMMARY:
This project will evaluate the impact of including Severe Combined Immunodeficiency into the newborn bloodspot screening panel. It will recruit parents and health professionals primarily from the sites where this new form of screening is being trialled well as additional sites where clinicians will be involved in the care of these babies and comparator groups are needed.

The proposed work will consist of two work packages. The first, a mixed-methods study conducted with families from the point of screening information being returned through to the child's fifth birthday. The second, a qualitative interview study conducted with health professionals during the clinical evaluation phase of the national pilot programme.

DETAILED DESCRIPTION:
BACKGROUND

Some countries have introduced newborn screening for Severe Combined Immunodeficiency (SCID) and modelling suggests it is probably cost effective in a UK setting. However, there is some uncertainty about this, and questions remain unanswered relating to its potential introduction in UK. The UK National Screening Committee (UKNSC) recommended that an evaluation should take place 'in practice' to try to answer some of these questions. The evaluation will take place in England and will involve about two thirds of babies born from September 2021 to August 2023. This amounts to approximately 800,000 newborns.

Screening for SCID within the NHS Newborn Blood Spot Screening Programme will make use of the blood spot already taken, usually by midwives, on babies at 5 days old. If, as a result of screening of this sample, babies are found to be at higher risk of SCID, parents will be notified, and the result explained. An appointment will be made for them to be seen the next day by an immunologist. At this appointment, the immunologist/clinical nurse specialist will explain the implications again and another blood test (flow cytometry) will be performed that day. The results are usually available the same day. These will be explained to the parent and depending on the result, they may be discharged ('false positive screening result') or appropriate management arranged ('true positive'). Amongst the true positives will be children with SCID, children who have other disorders (temporary or permanent) resulting in severe immune dysfunction and some children who have a problem with a particular part of their immune system (T cells) for whom the outcome is unknown on an individual basis. Although the target of the programme is SCID, children with the disorder are likely to represent only a minority of the true positives.

RATIONALE Previous research in other screening programmes has shown that delivering a false positive result to a participant, or asking them to attend hospital for further tests, following screening can have both short- and long-term deleterious effects. The size and nature of this in screening for SCID was one of the issues that the UKNSC wished to be explored. Preliminary survey and interview studies have started to explore the inherent communication dilemmas, the experiences of parents and health professionals. This project will seek to extend this work by exploring the views and experiences of parents and health professionals who participate in the clinical evaluation.

RESEARCH QUESTION/ AIMS

1. Family Study

   1. To explore the effects on families whose babies had a positive SCID screening test (low TRECs). This will include babies with normal results on confirmatory testing, as well as those with a result suggesting they have SCID or another disorder affecting their immune system.
   2. To compare views of the above families with families where the initial screening result did not put the child in a higher risk category and families who received a false positive result from another newborn bloodspot screening programme.
   3. To compare quality of life of children with SCID whose diagnosis was reached by screening, family history or symptomatic presentation.
   4. To measure the quality of life of families who have a child with secondary or syndromic T cell lymphopenia
   5. To measure the quality of life and screening experience of children with idiopathic T cell lymphopenia compared to experiences of families who have a child diagnosed with CFSPID.
2. Health Professional Study A) Explore the views and experiences of a sample of midwives who gained consent and took the initial blood sample.

B) To explore the views and experiences of the immunologists/clinical nurse specialists who saw the families at the time of flow cytometry.

N.B. Throughout this work we refer to 'parents' for simplicity. However, we recognise that the family situations of the infants may be more complex, with the existence of legal guardians and non-resident parents. The baseline position is for resident guardians to be included, but if specific circumstances suggest a wider parental group, additional participants may be included.

ELIGIBILITY:
Inclusion Criteria:

Participants must be at least 18 years of age. Participants must be able to understand the purpose and implications of the research study.

Where participants are speakers of languages other than English, the research team will arrange a translator.

Exclusion Criteria:

Where a child dies after recruitment to the project the team will sensitively check whether the parents wish to continue participation to enable their views to be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Parent Study A) Parents whose baby was referred to an immunologist due their SCID screening result B) Parents who received a normal screening result C) False positives elsewhere in screening D) Parents who received a CFSPID result E) Parents whose baby was identified with SCID due to family history or clinical presentation F) Parents who have received an abnormal screening result (T cell receptor excision circles (TRECs) or who were identified with SCID due to family history or clinical presentation and whose baby has subsequently died
  2. Health professional study Health professionals working in the evaluation centres will be invited to a semi-structured interview.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L, GAD-7, ITQOL-47 | Every 12 months until the child is 5 years of age
Qualitative interview data | Jan 2022-Sept 2023

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
TBC